CLINICAL TRIAL: NCT05552989
Title: Towards Better Preparedness for Future Catastrophes - a Qualitative Mixed Methods Study of Lessons Learned From Civil-military Disaster Response in Heidelberg, Germany, During the COVID-19 Pandemic
Brief Title: Towards Better Preparedness for Future Catastrophes - Local Lessons-learned From COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Markus Ries, MD PhD MHSc FCP, Professor, University Hospital Heidelberg
Other Study IDs: S-534/2022
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Pandemic; Emergencies
Keywords: COVID-19; disaster management; preparedness; lessons-learned; resilience
MeSH Terms: conditions — COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Key stakeholders of the local disaster relief community
  Interventions: Other: this is a non-interventional study

INTERVENTIONS:
Other: this is a non-interventional study — this is a non-interventional study

SUMMARY:
The research question of this study is: "what lessons have been learned from the civil-military cooperation in Heidelberg, Germany, during the COVID-19 pandemic, and what needs to be done to be better prepared for future disasters?" It is expected that the results of this research provide a deep expert insight into COVID-19 disaster preparedness at the local level. Flanked by comparison with published experiences at the global level, these lessons-learned would contribute to strengthening local crisis resilience sustainably in the future.

DETAILED DESCRIPTION:
Design, execution, analysis and publication of this study is conducted in compliance with the international quality criteria "STrengthening the Reporting of OBservational studies in Epidemiology (STROBE)" and "Standards for Reporting Qualitative Research (SRQR)".

This is a monocentric, qualitative, mixed-methods, non-interventional, non-randomized research project.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Direct or indirect involvement in civil-military collaboration during the COVID-19 crisis
3. Ability to provide consent
4. Providing written informed consent to participate in the study

Exclusion Criteria:

1) Failure to provide written informed consent to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Key stakeholders of the local disaster relief community
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Civil-military disaster relief support to Heidelberg, Germany, during the COVID-19 crisis | Years 2020 to 2022
  Autoethnographic qualitative, empiric-observational analysis
From civilian capability gaps towards societal resilience | One session of 2 hours (cross-sectional assessment at interview appointment)
  Structured interview with key stakeholders of the local disaster relief community
From lessons-learned towards better future disaster preparedness | One session of 2 hours (cross-sectional assessment at interview appointment)
  Structured interview with key stakeholders of the local disaster relief community

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ries, MD, PhD, MHSc, FCP, Principal Investigator — Heidelberg University
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schulze C, Welker A, Kuhn A, Schwertz R, Otto B, Moraldo L, Dentz U, Arends A, Welk E, Wendorff JJ, Koller H, Kuss D, Ries M. Public Health Leadership in a VUCA World Environment: Lessons Learned during the Regional Emergency Rollout of SARS-CoV-2 Vaccinations in Heidelberg, Germany, during the COVID-19 Pandemic. Vaccines (Basel). 2021 Aug 11;9(8):887. doi: 10.3390/vaccines9080887. PMID 34452012
- [Background] Ries M. Global key concepts of civil-military cooperation for disaster management in the COVID-19 pandemic-A qualitative phenomenological scoping review. Front Public Health. 2022 Sep 15;10:975667. doi: 10.3389/fpubh.2022.975667. eCollection 2022. PMID 36187698
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fpubh.2022.975667/full